CLINICAL TRIAL: NCT06141109
Title: Safety, Tolerability and Efficacy of MB07133 Plus Sintilimab in Patients With Hepatocellular Carcinoma，a Phase 1/2a Study
Brief Title: Treatment of MB07133 Plus Sintilimab in Patients With Hepatocellular Carcinoma
Acronym: MB07133
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Xintong Pharmaceutical Research Co.,Ltd. (Other)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H201110LC3
Record Dates: First submitted 2023-11-09; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Safety Issues; Efficacy; MTD
MeSH Terms: interventions — sintilimab; 4-amino-1-(5-O-(2-oxo-4-(4-pyridyl)-1,3,2-dioxaphosphorinan-2-yl)arabinofuranosyl)-2(1H)-pyrimidinone

STUDY DESIGN:
Intervention Model Description: MB07133 600mg/m2/day+Sintilimab 200mg、 MB07133 1200mg/m2/day+Sintilimab 200mg、 MB07133 1800mg/m2/day+Sintilimab 200mg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MB07133+Sintilimab (Experimental): The test is divided into 2 stages： fist stage is dose escalation：Sintilimab 200mg，MB07133 injection is divided into three dosage groups: 600mg/m2/day, 1200mg/m2/day, and 1800mg/m2/day.
  second stage Dose expansion：Sintilimab 200mg+MB07133 1800mg/m2/day
  Interventions: Drug: Sintilimab 200mg+MB07133 600mg

INTERVENTIONS:
Drug: Sintilimab 200mg+MB07133 600mg — 1. Adopting the classic "3+3" scheme design, 3 dose groups, with a cycle of 21 days. On the first day of each cycle, a single infusion of Sintilimab is given, and MB07133 is given for 7 consecutive days after a 2-hour interval between infusion initiation.
  2. Sintilimab 200mg+MB07133 1800mg, recruiting 30 subjects，the administration method is as 1.
  Other Names: Sintilimab 200mg+MB07133 1200mg; Sintilimab 200mg+MB07133 1800mg

SUMMARY:
An open-label, multi-dose clinical trial design was used to investigate the combination of MB07133 injection combined with Sintilimab in the treatment of primary liver cancer in phase I/IIa studies, including two phases of dose escalation and dose expansion，in order to evaluate the safety and efficacy of MB07133 injection combined with Sintilimab.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 70 years old (including 18 and 70 years old), regardless of gender;
2. Non resectable hepatocellular carcinoma/mixed liver cancer confirmed by pathological diagnosis (pathological tissue/cytology) or clinical diagnosis (dynamic enhanced MRI/dynamic enhanced CT scan);
3. At least one measurable lesion in the liver (in accordance with RECISIT1.1 standard);
4. Child-Pugh liver function score: A/B (≤ 7 points);
5. Expected survival time ≥ 12 weeks;
6. ECOG score of 0 or 1;
7. Patients who have completed chemotherapy/radiotherapy for tumors for more than 4 weeks (those who have received nitrosoureas and mitomycin chemotherapy for more than 6 weeks, those who have received small molecule targeted drugs (such as sorafenib and lovatinib) for more than 2 weeks), or those who have completed chemotherapy/radiotherapy for more than 5 half-lives (time limit whichever is longer), and those who have received the last intervention, radiotherapy, surgery, and ablation treatment for more than 4 weeks;
8. Not using any anti-tumor drugs within 2 weeks before the first medication;
9. Active hepatitis B patients should be controlled accordingly, and continue to take antiviral drugs and monitor liver function Can and hepatitis B virus load (such as: HBV DNA<104 copies/ml (2000IU/ml)).
10. If the main organ function is normal, it meets the following standards: blood routine examination: HGB ≥ 90 g/L; ANC ≥ 1.5 × 109/L; PLT ≥ 80 × 109/L; Blood biochemical test: ALB ≥ 28 g/L; ALT and AST ≤ 5.0 × ULNTBIL ≤ 1.5 × ULN; Creatinine ≤ 1.5 × ULN; The electrolyte is normal or normal after treatment or judged by the researcher to be abnormal without clinical significance; Urinary routine examination: Urinary protein ≤ 1+, if urinary protein ≥ 2+but 24-hour urinary protein<1.0g, it can be included in the group; ECG results: QTcB<470ms for males and<480ms for females; Thyroid function: Thyroid stimulating hormone (TSH) and free thyroxine (FT3) are within the normal range or have been determined by researchers to be abnormal without clinical significance.
11. Female patients of childbearing age or male patients with sexual partners of childbearing age should take effective contraceptive measures throughout the entire treatment period and 6 months after the last medication; Women of childbearing age cannot be in pregnancy or lactation.
12. The patient voluntarily signs a written informed consent form and is able to comply with the visit and related procedures stipulated in the plan.

Exclusion Criteria:

1. Moderate or higher amounts of chest/ascites and pericardial effusion with clinical symptoms; Those who have received chest/ascites drainage within the past month; Only a small amount of chest/ascites and pericardial effusion found on imaging without symptoms can be included in the group;
2. The main portal vein cancer thrombus simultaneously affects the contralateral portal vein branch, or simultaneously affects the superior mesenteric vein and inferior vena cava cancer thrombus, and has been confirmed by the researcher;
3. Previous history of liver transplantation;
4. Obstructive jaundice and liver failure, resulting in hepatic encephalopathy; Tumor invading the inferior vena cava and forming a tumor thrombus in the inferior vena cava; If histological/pathological results can be provided, patients with fibrous lamellar or sarcomatous hepatocellular carcinoma or cholangiocarcinoma cannot be included in the group;
5. Previous and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe damage to lung function, and other lung diseases;
6. Within 4 weeks before the first administration, immunosuppressive drugs have been used, excluding topical corticosteroids or physiological doses of systemic corticosteroids through nasal spray, inhalation, or other means. Temporary use of corticosteroids is allowed to prevent allergic reactions or treat respiratory distress symptoms such as asthma and chronic obstructive pulmonary disease;
7. Severe infections occurring within 4 weeks prior to the start of the study treatment, including but not limited to infection complications requiring hospitalization, bacteremia, severe pneumonia, etc;
8. Patients who have previously used immune checkpoint inhibitors (such as anti PD-1, anti PD-L1, and anti CTLA-4 antibodies) and have experienced the following immune checkpoint related adverse events, regardless of recovery, are not suitable for enrollment: a) ≥ Level 3 eye adverse events b) Level 4 liver dysfunction c) ≥ Level 3 neurological toxicity d) ≥ Level 3 colitis e) ≥ Level 3 renal toxicity f) ≥ Level 3 pulmonary inflammation;
9. For patients who receive radiation therapy 4 weeks before the first administration, all of the following conditions must be met before enrollment: currently, there are no toxic reactions related to radiation therapy, glucocorticoids do not need to be used, and radiation pneumonia, radiation hepatitis, radiation enteritis, etc. are excluded; Except for palliative radiotherapy for bone lesions within 7 days prior to the start of the study treatment;
10. HIV antibody positive individuals; Treponema pallidum specific antibody positive: if TRUST/RPR test is negative, it can be included in the group;
11. Active autoimmune diseases that require systemic treatment (such as the use of disease relieving drugs, corticosteroids, or immunosuppressants) have occurred within 2 years prior to the first administration. Allow the use of alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency). A known history of primary immunodeficiency. Patients with only positive autoimmune antibodies need to confirm the presence of autoimmune diseases based on the judgment of researchers;
12. Within 4 weeks before the first administration or planned to receive live attenuated vaccines during the study period;
13. Individuals with other primary malignant tumors within 5 years, except for non melanoma skin cancer and cervical cancer in situ that have received sufficient treatment;
14. Patients with active bleeding or abnormal coagulation function (PT>16s, APTT>43s, INR ≥ 2), bleeding tendency, or undergoing thrombolysis, anticoagulation, or antiplatelet therapy (excluding those who require heparin due to PICC or deep venous catheterization); Individuals with significant bleeding/loss of blood (greater than 450ml) within 28 days;
15. Simultaneously taking drugs (such as amiodarone, quinidine, etc.) that may prolong QTc and/or induce torsade de pointe (Tdp);
16. Pregnant or lactating women;
17. Any significant clinical and laboratory abnormalities that the researchers think affect the safety evaluation, such as: serious or medically important infections, uncontrolled diabetes (glycosylated hemoglobin>9.0%), patients with hypertension who cannot be reduced to the following range after treatment with two or less antihypertensive drugs (systolic pressure<160 mmHg, diastolic pressure<100 mmHg), peripheral neuropathy of grade II or above (CTC AE V5.0) Congestive heart failure, myocardial infarction within 6 months, etc.
18. History of hypertensive crisis or hypertensive encephalopathy;
19. Individuals with unstable central nervous system, meningeal metastasis, and mental disorders; Patients with stable brain metastasis after treatment (no need for treatment for at least 4 weeks) can be enrolled in the group;
20. Within the past 3 months, there has been a history of gastrointestinal bleeding or a clear tendency for gastrointestinal bleeding, such as known local active ulcer lesions;
21. Patients with significantly abnormal glomerular filtration rate;
22. Active hepatitis C, that is, those who are anti HCV positive and HCV RNA positive, and those who turn negative for HCV RNA after treatment can be included in the group; Individuals infected with acute or chronic hepatitis B or hepatitis C, with hepatitis B virus (HBV) DNA>2000IU/ml or 104 copies/ml; Hepatitis C virus (HCV) RNA>103 copies/ml; Hepatitis B surface antigen (HbsAg) and anti HCV antibody were positive at the same time.
23. After antiviral treatment, those who fall below the above standards can be enrolled in the group;
24. Active pulmonary tuberculosis (TB), who is receiving anti-tuberculosis treatment or has received anti-tuberculosis treatment within one year before the first administration;
25. Those who use any known drugs or substances that strongly inhibit or induce CYP3A4 liver microsomal enzymes 28 days prior to the use of the study drug ;
26. Subjects suspected to have a history of allergy to araC or similar drugs;
27. Symptoms of gout and blood uric acid>430 umol/L;
28. Any known deficiency in glutathione metabolism or the need for high doses of acetaminophen/Tylenol ® (>1 g/day), or subjects who require or use medication doses that will consume glutathione;
29. Patients who have participated in clinical trials of other drugs and used the study drug within 28 days prior to the use of the study drug (recorded as the last time the drug was used);
30. Subjects who the researchers believe have other factors that are not suitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with DLT Event | From initial administration to 21 days after starting administration
  According to the internationally recognized NCI-CTCAE 5.0 toxicity evaluation standard
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Starting to receive the experimental drug until 24 days after the last application
  All adverse medical events that occur after subjects receive the investigational product can be manifested as symptoms, signs, diseases, or laboratory abnormalities, but do not necessarily have a causal relationship with the investigational product.
PFS | Screening period, every 2 cycles after starting treatment（each cycle is 21 days）until the date of first documented progression or date of death from any cause（No more than 24 cycles are expected）.
  The time between the start of medication and the occurrence of objective tumor progression or death（RECIST1.1 ）

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) of Sintilimab | Within 0.5 hours before infusion，0.5hour (± 5 min) after the start of infusion，4hour(±5min)、10hour(±5min)、25hour(±30min)、73hour(±30min)、170hour.
  Pharmacokinetics of Sintilimab
Area Under the Plasma Concentration Versus Time Curve (AUC) of MB07133 | Within 0.5 hours before infusion，0.5hour (± 5 min) after the start of infusion，1hour(± 5min)、2hour(±5min)、4hour(±5min)、8hour(±5min)、12hour(±5min)、23hour(±30min)、 47hour(±30min)、71hour(±30min)、119hour(±30min)、143hour(±30min)、168hour
  Pharmacokinetics of MB07133

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Jilin, Changchun, China